CLINICAL TRIAL: NCT04543851
Title: CARA Treatment Pilot Study for Breast Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Cheryl Duzenli, Medical Physicist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H18-02014
Record Dates: First submitted 2020-08-25; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Side Effect
Keywords: skin dose; skin fold; organ at risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CARA positioning (Experimental): Planning and Treatment using the CARA Device
  Interventions: Device: CARA - carbon fibre adjustable re-usable accessory for breast positioning

INTERVENTIONS:
Device: CARA - carbon fibre adjustable re-usable accessory for breast positioning — Breast positioning to alleviate infra-mammary fold and lateral breast sag

SUMMARY:
CARA is a novel Carbon-fibre Adjustable and Re-usable Accessory for supine breast positioning during radiation therapy. CARA was developed at BC Cancer. In this study, twenty patients will be planned and treated with CARA positioning to establish safety and workflow measures of this novel device. The device is designed to remove the infra-mammary skin fold and lateral breast droop which can lead to unwanted dose to normal tissue.

DETAILED DESCRIPTION:
This pilot study will investigate the safety and potential benefits of CARA breast positioning by treating 20 patients using the device. Patients will be planned with CARA positioning and standard of care positioning. CARA plans will be evaluated to ensure all treatment planning goals are met and patients will proceed to treatment with CARA positioning. This pilot study will ensure that patients can be safely treated with the CARA and provide us with valuable information from therapists, oncologists and patients about the performance of the current design. This will also inform the direction of design improvements and the production of educational materials for training practitioners in the use of the device. Overall, this will prepare us for a randomized clinical trial of the CARA positioning technique versus current standard of practice to assess whether reduced toxicity can be achieved using the CARA technique.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with completely excised stage I or II invasive breast cancer, or ductal carcinoma in situ (DCIS), who have undergone breast-conserving surgery and are scheduled to undergo adjuvant breast radiotherapy;

Any breast size with a skin fold of depth 1 cm or greater at the infra-mammary crease at the time of radiation treatment planning, or brassiere cup size equal to or larger than D;

Patients undergoing nodal radiotherapy are eligible if the above criteria are met;

Patients undergoing boost radiotherapy are eligible if the above criteria are met, but only if the surgical scar does not extend inferior to the nipple line of the breast;

Language is not a barrier if there are interpreters/family members to translate;

Patients having had chemotherapy are eligible for this study;

Exclusion Criteria:

Inability to give informed consent or comply with requirements of the trial;

Failure of healing of the surgical scar or significant post-operative wound infection;

Prior radiotherapy to either breast or to the chest;

Presence of significant connective tissue disease (e.g. systemic sclerosis); known radiation hypersensitivity phenotype (e.g. ataxia telangiectasia);

Inability to return for assessment at both one week and two weeks following completion of radiotherapy;

Breast reconstruction;

Use of Mepitel® wound dressing product.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Number of participants for whom dose volume treatment planning constraints are not met using CARA support for breast setup | 12 months
  Treatment planning dose constraints are:
  >=95% of the prescribed dose covering >=98% of the breast target tissue, including internal mammary chain when requested by the treating oncologist
  volume of ipsi-lateral lung receiving >= 20Gy should be <=35%
  volume of heart receiving >=25Gy should be <=5%
  maximum dose to any point in the body <=110% of the prescribed dose
  volume of breast receiving >=107% of prescribed dose should be <=22 cm^3
Number of participants having measured breast skin dose => 110% of the prescribed dose to an area of skin => 1 cm^2 | 12 months
  Skin dose is measured on the breast surface under the carbon fibre device using radio-chromic film. The area of skin receiving 70% of the prescribed dose up to the maximum absorbed dose is measured in 5% dose increments to an accuracy of 0.5 cm^2.
  If any participant receives => 110% of the prescribed dose to >=1 cm^2 area of skin, the study will be stopped.
Number of participants scoring =>6 on the CTCAE Version 4.0 skin assessment | 12 months
  Participants will undergo a detailed breast skin assessment at baseline, one week prior to RT completion, last week of RT, and one and two weeks post RT using the CTCAE Version 4 skin assessment scoring system as well as examination of the infra-mammary fold for any moist desquamation. The dimensions and location of moist desquamation will be recorded. In the event that a skin reaction of ≥ 6 (indicating ulceration, hemorrhage or necrosis) on the CTCAE V 4.0 scale is reported, the trial will be stopped.

SECONDARY OUTCOMES:
Workflow measures | 12 months
  Measured time to accomplish set up and treatment with CARA positioning
Setup reproducability | 12 months
  Measure required shifts in patient position using kilo-voltage imaging
Doses to organs at risk comparison with standard of care | 12 months
  Comparison of lung, heart, breast and normal tissue dose versus standard of care
Skin assessment versus skin dose | 12 months
  CTCAE V4 and specific moist desquamation assessment of breast skin compared with measured skin dose-area data
Patient Reported outcome - skin reaction | 12 months
  Questionnaire to assess patient reported side effects and skin reaction

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl R Duzenli, PhD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malhotra A, Chan EK, Nichol A, Duzenli C. Spatial dose-distribution-based risk mapping to predict moist desquamation in breast radiotherapy. Phys Med Biol. 2025 May 27;70(11). doi: 10.1088/1361-6560/add985. PMID 40373801
- [Derived] Duzenli C, Koulis T, Menna T, Carpentier E, Arora T, Coope R, Gill B, Lim P, Aquino-Parsons C, Nichol A, Singer J, Ingledew PA, Grahame S, Chan EK. Reduction in Doses to Organs at Risk and Normal Tissue During Breast Radiation Therapy With a Carbon-Fiber Adjustable Reusable Accessory. Pract Radiat Oncol. 2021 Nov-Dec;11(6):470-479. doi: 10.1016/j.prro.2021.06.012. Epub 2021 Jul 21. PMID 34303034